CLINICAL TRIAL: NCT05086575
Title: Observatory of Patients With Haemophilia B Treated by IdElvion®
Acronym: OrPHEe
Status: Active, not recruiting | Type: Observational
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Other Study IDs: OrPHEe study; 2021-A00468-33 (Other: ANSM)
Record Dates: First submitted 2021-09-28; First posted 2021-10-21 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Haemophilia B
Keywords: FIX, Coagulation FIX
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
OrPHEe is a non-interventional, prospective and national study which aim is to record real life data in haemophilia B French patients treated with Idelvion® to confirm the efficacy and safety of this product established in clinical development studies.

DETAILED DESCRIPTION:
Haemophilia B is a congenital coagulation disorder caused by a deficiency or anomaly of coagulation factor IX (FIX).

The severity of the haemophilia depends on the extent of the FIX deficiency with clinical manifestations differing depending on the location of the bleed.

Treatment of this disease involves the administration of the deficient factor, i.e. FIX, to patients. Depending on the severity of the disease and context, a range of treatment regimens are available (long-term prophylactic treatment for the prevention of non-surgical bleeds, short-term prophylactic treatment for high-risk periods, treatment for the prevention of surgical bleeds or on-demand curative treatment).

CSL Behring has developed a long-acting recombinant FIX, i.e. rIX-FP (Idelvion®), to extend the intervals between the administrations of treatment while also providing a therapeutic benefit. Data from clinical studies clearly confirm the therapeutic benefit of Idelvion® in adult and paediatric patients with haemophilia B previously receiving an on-demand treatment for bleeding episodes, for long-term prophylaxis, as well as in patients undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* Have agreed to participate in the observatory after receiving written information on the purpose of the study and the personal data to be collected (agreement of parents for under-age patients);
* Present with haemophilia B and are currently being treated or have previously been treated with Idelvion® as a long-term prophylactic treatment, on-demand treatment or short-term treatment for surgical procedures or to cover periods with a high-risk of bleeding.
* Do not have FIX targeted antibodies at the time of the inclusion visit

Exclusion Criteria:

* Refusal by the patient or his/her legal representative to participate in the study;
* Existence of a contraindication to the use of Idelvion® treatment (known hypersensitivity to FIX or hamster proteins);
* Simultaneous participation in an interventional clinical study on a drug

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Haemophilia B patients treated with Idelvion®
Sampling Method: Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Annual bleeding rates (overall, spontaneous and traumatic) under the scope of long-term prophylaxis or on-demand treatment of non-surgical bleeding events | Up to 36 months
Number of spontaneous bleeding events per patient | Up to 36 months
Number of Idelvion® infusions and doses injected by infusion required to prevent and resolve non-surgical bleeding episodes | Up to 36 months
Incidence of non-surgical bleeding episodes | Up to 36 months

SECONDARY OUTCOMES:
The number of infusions and total dose of Idelvion® (in IU/kg) required to prevent or treat surgical bleeding episodes | up to 36 months
Incidence of surgical bleeding episodes | up to 36 months
The number of infusions and total dose of Idelvion® (in IU/kg) required to cover a high risk of bleeding | up to 36 months
The number of infusions and total dose of Factor IX consumed in the year prior to taking Idelvion® | up to 36 months
The number of infusions and total dose of Idelvion® | up to 36 months
The type and incidence of adverse events (AE) in particular severe AE,and AE related to Idelvion® | up to 36 months
Completion of the following questionnaire: EQ-5D-3L for adults | up to 36 months
Completion of the following questionnaire: EQ-5D-Y for children from 8 to 12 years | up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Catovic, Study Director — CSL Behring SA
Locations (28):
- France (28):
  - CHU Amiens - Picardie, Amiens
  - CH Annecy Genevois, Annecy
  - CHRU Besançon, Besançon
  - CHU Bordeaux - Hôpital Pellegrin, Bordeaux
  - CHRU Brest, Brest
  - CHU Caen, Caen
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Dijon, Dijon
  - Hôpital Simone Veil, Eaubonne
  - CHU de Grenoble, Grenoble
  - CRC-MHC Hôpital Kremlin Bicêtre, Le Kremlin-Bicêtre
  - CH du Mans, Le Mans
  - CHRU Lille, Lille
  - CHU de Limoges, Limoges
  - Hôpital Edouard Herriot, Lyon
  - CHU Montpellier, Montpellier
  - CHRU Nancy, Nancy
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - Hôpital Necker Enfants Malades, Paris
  - CHU de Reims, Reims
  - CHU Rennes, Rennes
  - CHU Rouen, Rouen
  - CHU Saint-Etienne, Saint-Etienne
  - CHRU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours
  - Hôpital André Mignot - CH Versailles, Versailles